CLINICAL TRIAL: NCT01193075
Title: Natural History Evaluation of Charcot Marie Tooth Disease (CMT) Type (CMT1B), 2A (CMT2A), 4A (CMT4A), 4C (CMT4C), and Others
Brief Title: Natural History Evaluation of Charcot Marie Tooth Disease (CMT) Types CMT1B, CMT2A, CMT4A, CMT4C, and Others
Acronym: INC-6601
Status: Recruiting | Type: Observational
Sponsor: Michael Shy (Other)
Collaborators: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Johns Hopkins University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); King's College Hospital NHS Trust (Other); Nemours Children's Hospital (Other); Stanford University (Other); University of Pennsylvania (Other); University of Rochester (Other); Children's Hospital of Philadelphia (Other); Sydney Children's Hospitals Network (Other); Rare Diseases Clinical Research Network (Network); Muscular Dystrophy Association (Other); National Institutes of Health (NIH) (NIH); Charcot-Marie-Tooth Association (Other); Massachusetts General Hospital (Other); Cedars-Sinai Medical Center (Other); University of Miami (Other); University of Minnesota (Other); Connecticut Children's Medical Center (Other); University of Colorado, Denver (Other); The National Hospital for Neurology and Neurosurgery (Unknown); Dubowitz Neuromuscular Centre (Other)
Responsible Party: Sponsor-Investigator, Michael Shy, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: INC-6601; 1U54NS065712-01 (NIH)
Record Dates: First submitted 2010-08-09; First posted 2010-09-01 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2024-05

CONDITIONS: Charcot Marie Tooth Disease
Keywords: Charcot Marie Tooth disease; CMT; HMSN; HMN; HSN; CMT1; CMT2
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Hereditary Sensory and Motor Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- CMT1B: Families/patients with genetically confirmed CMT1B
- CMT2A: Families/patients with genetically confirmed CMT2A
- CMT4A: Families/patients with genetically confirmed CMT4A
- CMT4C: Families/patients with genetically confirmed CMT4C
- All other CMT: Families/patients with all other forms of CMT or CMT that has not yet been genetically identified

SUMMARY:
This is an observational longitudinal study to determine the natural history and genotype-phenotype correlations of disease causing mutations in Charcot Marie Tooth disease (CMT) type 1B (CMT1B), 2A (CMT2A), 4A (CMT4A), and 4C (CMT4C).

The investigators will also be determine the capability of the newly developed CMT Pediatric Scale (CMT Peds scale) and the Minimal Dataset to measure impairment and perform longitudinal measurements in patients with multiple forms of CMT over a five year window

DETAILED DESCRIPTION:
The Inherited Neuropathies Consortium (INC) is a member of the Rare Disease Clinical Research Network (RDCRN) that is funded by the National Institutes of Health (NIH) through the Office of Rare Diseases (ORD) and the NINDS. The University of Iowa is the lead center in INC which also includes sites from the University of Pennsylvania, Children's Hospital of Philadelphia (CHOP), the University of Rochester (NY), the National Hospital for Neurology and Neurosurgery in London England, the Dubowicz Neuromuscular Center, and the University of Miami (Florida). The North American CMT Network is an additional consortium that is funded by the Muscular Dystrophy Association (MDA) and the Charcot Marie Tooth Association (CMTA). The University of Iowa is the lead site for this consortium as well. Additional sites include the University of Washington (Seattle), Vanderbilt University, Johns Hopkins University, the University of Sydney, the Besta Neurological Institute in Milan (Italy), Harvard University and the intramural Neurogenetics division of the NIH. All funding sources have agreed to allow us to house data from the two consortia together at the NIH funded Data Management Coordinating Center (DMCC) at the University of South Florida and to group them under the name of the Inherited Neuropathies Consortium (INC).

The inherited peripheral neuropathies are often called Charcot Marie Tooth Disease (CMT), named after the three physician scientists who first described them. These are a heterogenous group of disorders caused by mutations in more than 50 different genes. The diseases cause weakness and loss of sensation in patients. There are no effective treatments for any forms of CMT. There is also limited information on the natural history of how any of the different types of CMT progress and limited outcome measures to measure impairment. The purpose of INC is to investigate the natural history of the different types of CMT, to identify genes that modify the severity of individual types of CMT, to develop and test outcome measures for children with CMT, to develop an interactive website for patients with CMT and to develop the knowledge needed to perform clinical trials in patients with CMT.

To do this, people who have, are suspected to have, or have a family history of an inherited neuropathy will take part in a full-day evaluation. These patients are being seen in order to receive a possible diagnosis of CMT and clinical care, but may also choose to participate in this research project. Most of the testing being performed would be done as part of the standard of care for diagnosing and treating a patient with an inherited neuropathy. Additional testing may be performed on certain subjects if applicable, but the majority of subjects who volunteer for this study are allowing us to use the clinical information obtained during their visit as coded data for natural history purposes and to develop outcome measures.

Because all individuals who attend the CMT clinic would be eligible for participation in this study, when they arrive for their clinic visit, the initial meeting is to review the consent form for the research project. Thus, the evaluation will begin with consenting subjects into the study, if applicable. Then, a variety of tests will take place to measure the presence and severity of symptoms, along with identifying which type of CMT a patient/subject may have. Tests included in this study which are also the standard of care for patients with inherited neuropathies include a neurological evaluation by a trained neurologist, a limited set of nerve conduction studies, physical therapy assessment, orthotist assessment, genetic counseling, and possibly genetic testing to determine the form of CMT. Additional clinical testing which may be used for research includes EMGs or MUNE testing to evaluate possible muscular dystrophies or muscle involvement in the disease. The results from these tests will be used for diagnostic purposes and to give each patient a CMT Neuropathy Score (CMTNS) which is a validated instrument that allows us to assess the severity of disease based on a 36 point scale. If the subject is also involved in the research project, the results will also be used for research purposes.

Additionally, some subjects may undergo testing which is not a part of regular clinical care, but is being done for research purposes only. These tests/procedures may include hand function testing, physical assessment using the CMT Peds Score (an instrument used to evaluate children with CMT - see substudy 6603), research based genetic testing, quality of life questionnaires, or a skin biopsy. All of these tests/procedures are optional, subjects do not have to complete these to be involved in the overall natural history study. Opting out of any of these procedures does not mean that they would be excluded from the study. Some of these procedures would only be performed on certain individuals who are eligible based on age or type of CMT. Skin biopsies are being performed on certain qualified subjects for research purposes in order to grow fibroblast cells to further study various forms of CMT. These individuals would be over 18 and have specific forms of CMT.

Additionally, there are sub-studies that are being performed which SOME subjects may be eligible for. These sub-study options will be discussed with each patient prior to their participation.

Sub-study #6601 - Test-retest protocol addendum for pCMT-QOL. Substudy for a small group of subjects in order to assess the test-retest reliability indicates reproducibility of the pCMT-QOL. In order to calculate test-retest reliability, at a single site of the Inherited Neuropathy Consortium (University of Iowa), 25 subjects aged 8-18 and their parents will be given the appropriate version of pCMT-QOL, as well as the parents of 10 subjects aged 7 and under. These parents will in addition be given a pre-stamped envelope containing the same version of the pCMT-QOL that they took, to be completed by their child and/or parent in 4 weeks and return by mail (in CMT, the disease should not fluctuate in a 4 week interval). Parents will be given one reminder phone call in 6-8 weeks, and the pCMT-QOL forms will be mailed to them again if they are reported missing. Test-retest reliability will be estimated by intraclass correlation coefficients (two-way random effects model) to show correlations between any given individual's scores in two QOL assessments taken 4 weeks apart.

Sub-study #6602 - This project is to understand modifier genes and how they influence the severity of disease expression, along with identifying new forms of CMT which have not been genetically determined. Subjects who are eligible will either have CMT type 1A (CMT1A) or an unknown form of CMT type 2 (CMT2). Blood will be drawn and sent to the University of Miami where they receive the coded sample and process it through exome sequencing. Subjects will be told that this is optional.

Sub-study #6603 - This project is to develop a new CMT Pediatric Scale (CMT Peds) for Children with CMT. Although there is a validated score (the CMTNS) which measures disease severity for CMT, it is not always applicable to children due to their limited ability to relay information about their symptoms. The CMT Peds scale is being developed and validated in order to measure disease severity in children and have outcome measures available for future clinical trials. Children (defined as 21 and under) being evaluated will be asked to perform functional tasks such as using stairs, walking in a hallway, and performing hand function tests. This information will be used to validate the CMT Peds score. Subjects will be informed that this study is optional.

These tests will be performed in one day during the clinic visit. Patients who attend the clinic are given the option of returning for annual visits to help with disease management. If a patient decides to follow up in the clinic, they will once again be asked to participate in the research. They do not need to participate in the research in order to be seen in the clinic, and they can opt out at any time. If a subject does not follow up by making an appointment in the clinic, they will not be contacted by us to schedule a return visit. All return visits are initiated by the patient/subject. An individual can decide not to participate in the research, but will still be able to be seen in the clinic and receive medical recommendations, treatment, and care by the clinical team who specializes in inherited neuropathies.

ELIGIBILITY:
Inclusion Criteria:

All patients must be seen in-person at a participating center for the initial visit.

Inclusion Criteria - patients with CMT (all subtypes)

1. Patient has documented, pathogenic or likely pathogenic CMT-causing variant(s)

   OR
2. Patient has a first- or second-degree family member (parent, child, sibling, half-sibling, aunt, uncle, grandparent, or grandchild) with a documented pathogenic or likely pathogenic CMT-causing variant AND a clear link between that family member and the affected patient AND a phenotype consistent with the diagnosis

   i. A clear link is necessary for a second-degree relative. For example, if a grandparent is affected and has a pathogenic or likely pathogenic variant, and the parent does not have any signs, symptoms, or electrophysiology consistent with the diagnosis, there is no clear link unless the parent has also been found to have the pathogenic or likely pathogenic variant such as in cases with reduced penetrance

   ii. In cases where clear links are not available, genetic testing is required for the patient or the family member who is not clearly affected.
3. Patients who have a variant of uncertain significance, as determined by the laboratory performing the testing may still be included if one of the following circumstances applies:

   i. Variant is categorized as pathogenic or likely pathogenic per the ACMG variant interpretation guidelines. [80, 81]

   ii. Variant has been found in multiple affected people in a family and has not been found in unaffected family members. (Note - both affected and unaffected family members must be tested in this situation to be included).

   iii. The principal investigator and the site investigator agree that the variant(s) is (are) most likely pathogenic.
4. Patients whose clinical presentation is suggestive of CMT, but CMT type and variant are unknown will be characterized by the following categories:

   1. Nerve conduction velocities: demyelinating, axonal, intermediate
   2. Inheritance: dominant, recessive, X-linked, or unknown
5. Patient or patient's legally authorized representative has understood and signed an IRB approved consent form for the study. Teenagers (age 13 - 17 years) and cognitively impaired adults who are able to read and write must sign an assent form (depending on local ethics committee requirements).

Inclusion Criteria - Controls

1. Person does not have a peripheral neuropathy, as determined by the investigator.
2. Person has understood and signed an IRB approved consent form for the study. Teenagers (age 13-17 years) must sign an assent form (depending on local ethics committee requirements).

EXCLUSION CRITERIA

1. Patient has a variant of uncertain significance that cannot be further classified following methods listed in the Inclusion Criteria.
2. Patient does not wish to be a part of the study or has not signed an informed consent form.
3. Patient is deemed inappropriate by the Site PI.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who present to a participating site and have Charcot Marie Tooth disease (CMT) will be recruited for participation.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Charcot Marie Tooth Neuropathy Score (CMTNS) | 1 year
  Charcot Marie Tooth Neuropathy Score (CMTNS) is a composite measure of disability based on a person's symptoms, signs, and electrophysiology. It is based on a 36 point scale, with 9 items each worth up to 4 points. A higher score signifies increased disability.
Minimal dataset | 1 year
  This includes diagnosis, family history, developmental history, walking ability, hand function, strength, sensation, and neurophysiology.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Shy, MD, Principal Investigator — University of Iowa
Locations (22):
- United States (18):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Connecticut/Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Nemours Children's Health, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard/Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Rochester, Rochester, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Children's Hospital, Seattle, Washington
- University of Westmead, Sydney, New South Wales, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- C. Besta Neurological Institute, Milan, Milan, Italy
- National Hospital of Neurology and Neurosurgery, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified RDCRN data is submitted to an ORDR-designated repository. For the current grant cycle, that repository has been dbGaP.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For Observational/Longitudinal/Natural History/Epidemiology studies): For the current grant cycle, available data will be released to the repository and will become available to the scientific community one year after publication of planned analyses, or after a period of 5 years from the date when the data were collected, whichever comes first.
Access Criteria: - For the current grant cycle, once de-identified data is posted on dbGaP, a summary of the study is posted and individual participant data is accessed via a request through dbGaP.
URL: https://www.ncbi.nlm.nih.gov/gap

REFERENCES:
- [Derived] Fridman V, Sillau S, Acsadi G, Bacon C, Dooley K, Burns J, Day J, Feely S, Finkel RS, Grider T, Gutmann L, Herrmann DN, Kirk CA, Knause SA, Laura M, Lewis RA, Li J, Lloyd TE, Moroni I, Muntoni F, Pagliano E, Pisciotta C, Piscosquito G, Ramchandren S, Saporta M, Sadjadi R, Shy RR, Siskind CE, Sumner CJ, Walk D, Wilcox J, Yum SW, Zuchner S, Scherer SS, Pareyson D, Reilly MM, Shy ME; Inherited Neuropathies Consortium-Rare Diseases Clinical Research Network (INC-RDCRN). A longitudinal study of CMT1A using Rasch analysis based CMT neuropathy and examination scores. Neurology. 2020 Mar 3;94(9):e884-e896. doi: 10.1212/WNL.0000000000009035. Epub 2020 Feb 11. PMID 32047073
- [Derived] Panosyan FB, Laura M, Rossor AM, Pisciotta C, Piscosquito G, Burns J, Li J, Yum SW, Lewis RA, Day J, Horvath R, Herrmann DN, Shy ME, Pareyson D, Reilly MM, Scherer SS; Inherited Neuropathies Consortium-Rare Diseases Clinical Research Network (INC-RDCRN). Cross-sectional analysis of a large cohort with X-linked Charcot-Marie-Tooth disease (CMTX1). Neurology. 2017 Aug 29;89(9):927-935. doi: 10.1212/WNL.0000000000004296. Epub 2017 Aug 2. PMID 28768847
- [Derived] Fridman V, Bundy B, Reilly MM, Pareyson D, Bacon C, Burns J, Day J, Feely S, Finkel RS, Grider T, Kirk CA, Herrmann DN, Laura M, Li J, Lloyd T, Sumner CJ, Muntoni F, Piscosquito G, Ramchandren S, Shy R, Siskind CE, Yum SW, Moroni I, Pagliano E, Zuchner S, Scherer SS, Shy ME; Inherited Neuropathies Consortium. CMT subtypes and disease burden in patients enrolled in the Inherited Neuropathies Consortium natural history study: a cross-sectional analysis. J Neurol Neurosurg Psychiatry. 2015 Aug;86(8):873-8. doi: 10.1136/jnnp-2014-308826. Epub 2014 Nov 27. PMID 25430934
- See also: Inherited Neuropathies Consortium Website — https://www.rarediseasesnetwork.org/cms/INC